CLINICAL TRIAL: NCT02304939
Title: Prospective, Randomized, Multi-center Trial Aiming to Determined the Impact of Changeovers of Norepinephrine on the Blood Pressure Stability With Patients in Shock in ICU.
Brief Title: CHangeovers of Norepinephrine in Intensive Care
Acronym: CHIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHRIP-2013; 2014-A00591-46 (Other: ID RCB)
Record Dates: First submitted 2014-11-24; First posted 2014-12-02 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Shock; Intensive Care
Keywords: Norepinephrine; Intensive Care; Changeovers; Smart pumps; Quick change; Double pumping; Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Quick change (Active Comparator): For this changeover : When the syringe of norepinephrine stops (pre alarm), start the second syringe pumps at the same speed of the first, wait for a first drop at the end of the tubing.
  Close the first syringe, disconnect it and connect the second syringe, open the valve on and stop the first syringe.
  Interventions: Procedure: changeover; Behavioral: datas collection
- Double Pumping (Experimental): For this changeover : When the syringe of norepinephrine stops (pre alarm), start the second syringe pumps, open the second syringe while leaving the first syringe open. Wait until the blood pressure rises 5 mmHg (SBP, DBP or MAP).
  Once the blood pressure increased or 2 minutes from the start of the relay if no increase in blood pressure is observed, close the first syringe.
  Interventions: Procedure: changeover; Behavioral: datas collection
- Smart infusion pump (Experimental): For this automatic changeover : When the syringe of norepinephrine stops (pre alarm), oversee the progress of the automatic relay.
  Interventions: Procedure: changeover; Device: use of automatic infusion pump; Behavioral: datas collection

INTERVENTIONS:
Procedure: changeover
Device: use of automatic infusion pump
  Arms: Smart infusion pump
Behavioral: datas collection

SUMMARY:
CHIC study's purpose is to compare the efficiency, in terms of blood pressure stability, of three changeovers of norepinephrine used routinely in ICU. The three techniques are:

* Quick change
* Double pumping
* Smart infusion pumps

DETAILED DESCRIPTION:
The drugs used in intensive care units are numerous and their administration is based on a strong expertise in this context of urgency and complexity. Nurses role is not only to carry out preparation of a treatment but to implement a complex treatment that requires a risk management approach surpassing the simple task to which the decree of professional acts refers to.

In this context, the administration of catecholamines, widely used in intensive care medicine in the treatment of shock, appears to be a sensitive issue to study. These vasoactive drugs have a short half-life and a narrow therapeutic index. Administration should be careful ensuring both efficiency and prevention of complications such as hemodynamic instability or arrhythmias.

Administration of these therapeutic must be strictly continuous, that is to say delivered using electric syringe pumps. Syringe replacements appear as critical moments because of the risk of flow change or brief interruption of the infusion.

There are three main types of syringes relay techniques, but to date, no study has compared these techniques with each other. There is thus no recommendation based on objective datas to guide clinical nursing practice.

This study aims to provide evidence in order to secure the administration of catecholamines. It may also use as a reference for evaluation of new features that allow automation relays with called "smart pumps" and for which no study has demonstrated the added value in terms of security. No progress will be possible in securing the administration of drugs with a short half-life, narrow therapeutic index and significant side effects without a deep reflection of the conditions of their infusion. The choice of materials used and the development of care procedures must be based on reliable and timely recommendations. Patients expect safer care. Nurses must be able to have references enabling them to guide their practice to the benefit of patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission in Intensive Care Unit
* Norepinephrine perfusion started for less than three hours in ICU
* Invasive monitoring of blood pressure

Exclusion Criteria:

* Age under 18
* Pregnant and breastfeeding women
* Previous participation in the trial
* No registration in any health care system
* Patient protected by law
* Patient study refusal
* Active therapeutic limitation decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
percentage of norepinephrine' syringes causing a change in the mean blood pressure over 15 mmHg | in the 15 minutes following the beginning of the relay

SECONDARY OUTCOMES:
Percentage of norepinephrine syringe's relays causing a hypotension defined by a 15 mmHg decrease of the mean blood pressure | in the 15 minutes following the beginning of the relay
Percentage of norepinephrine syringe's relays causing a hypertension defined by a 15 mmHg increase of the mean blood pressure | in the 15 minutes following the beginning of the relay
Average time in minute spend by a nurse to change the syringe | 15 minutes following the beginning of the relay

CONTACTS AND LOCATIONS:
Locations (1):
- Le Roy, Angers, France

REFERENCES:
- [Derived] Poiroux L, Le Roy C, Ramelet AS, Le Brazic M, Messager L, Gressent A, Alcourt Y, Haubertin C, Hamel JF, Piquilloud L, Mercat A. Minimising haemodynamic lability during changeover of syringes infusing norepinephrine in adult critical care patients: a multicentre randomised controlled trial. Br J Anaesth. 2020 Oct;125(4):622-628. doi: 10.1016/j.bja.2020.06.041. Epub 2020 Jul 29. PMID 32739045